CLINICAL TRIAL: NCT06772883
Title: The Effect of Sexual Education-Counseling According to PLISSIT in Solving Sexual Problems in Women Using Contraceptive Methods: One Year Follow-up Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Özlem BAKAN DEMİREL, PhDc, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARMARAU-SBE-OBD-02
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Contraception; Female Sexual Function; Sexual Dysfunction; PLISSIT; Training-consulting
Keywords: contraception; female sexual function; sexual dysfunction; PLISSIT; training-consulting
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Counseling; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental : Participant Group (Experimental): The women included in the Working Group were contacted by phone and invited to the hospital. Sexual education and counseling were provided in accordance with the PLISSIT model. A total of 5 interviews were conducted with the women, the first face-to-face interview and the subsequent ones by telephone. FSFI assessments in the study FSFI assessments were performed 5 times (initial, 1st, 3rd, 6th months and 1 year later). According to the PLISSIT model, their sexuality and any problems since the previous assessment were discussed and a short counseling was given if necessary.
  Interventions: Behavioral: sexual education and counseling
- Control Group (Other): Routine clinical care
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: sexual education and counseling — The women included in the Working Group were contacted by phone and invited to the hospital. Sexual education and counseling were provided in accordance with the PLISSIT model. A total of 5 interviews were conducted with the women, the first face-to-face interview and the subsequent ones by telephone. FSFI assessments in the study FSFI assessments were performed 5 times (initial, 1st, 3rd, 6th months and 1 year later). According to the PLISSIT model, their sexuality and any problems since the previous assessment were discussed and a short counseling was given if necessary.
  Arms: Experimental : Participant Group
Other: control group — routine clinical care
  Arms: Control Group

SUMMARY:
Sexuality is a universal part of human life and is a process in which two people share their emotions, body, soul and pleasures. Although it is a natural part of life, sexuality can be affected by many factors. One of these factors is the contraceptive methods used by couples. While contraceptive methods prevent unplanned/unwanted pregnancies and help couples to have a satisfying sexual life without the fear of becoming pregnant, they can also negatively affect the sexuality of couples and even cause sexual dysfunctions.

DETAILED DESCRIPTION:
Although there are many studies in the literature examining the changes of contraceptive methods on sexual behaviors, the relationship between method use and female sexual function remains unclear. There are studies showing that contraceptive method use has negative effects on sexual function (decreased frequency of sexual intercourse, difficulty in arousal, orgasm or lubrication), as well as studies suggesting that it may improve sexual behaviors. Some studies report that the contraceptive method used has no effect on sexual function.In contraceptive counseling, it is important to evaluate the sexual functions of the applicant and provide sexual counseling when necessary. It is recommended that health professionals use a model to effectively evaluate sexual functions and provide the most appropriate care in the presence of CD. In this direction, the education-counseling provided with the PLISSIT model, which is frequently used in this direction, can be an approach that can bridge the gap between the health professional and the individual in the elimination of CD.There are studies showing that sexual education-counseling using this model is effective. However, the number of studies in the literature in which the PLISSIT model was used to solve the problems of women experiencing CD during contraceptive method use is very limited. In addition, there is no study evaluating the effectiveness of the training-counseling provided with this model for 1 year in the literature. With the aim of contributing to the literature in line with this need, this study aimed to examine the effect of sexual education-counseling given in line with the PLISSIT model on the solution of sexual problems in women using contraceptive methods in a one-year period.

ELIGIBILITY:
Inclusion Criteria:

* ≤45 years of age and not in the peri/postmenopausal period (not menopausal which is),
* Has a sexual partner and has an active sexual life,
* One of the effective contraceptive methods (IUD, COC, Condom; Injection method, implanaon) for ≥3 months,
* Turkish language is not a problem,
* Educated enough to understand what they read and answer questions,
* Chronic diseases that may affect sexual health (cancer, diabetes, hypertension, hypercholesterolemia, heart disease, atherosclerosis, chronic pulmonary and hepatic diseases, chronic renal failure, etc.) or medication (antihypertensive, diuretic, lipid-lowering agent, H2 receptor antagonist, antihistamine, anticholinergic, chemotherapeutic agent, anticonvulsant, antidepressant, antipsychotic, narcotic, sedative) with no use and
* Women who volunteered to participate in the study were included in the study sample.

Exclusion Criteria:

* Applying for the first time/to use a new method,
* ≥46 years of age or menopausal,
* New to their current method (<3 months),
* Those who do not have an active sex life or who have very infrequent sex due to their partner's job, etc. in a relationship,
* Chronic illness or medication that may affect sexuality,
* Who doesn't speak Turkish,
* Not educated enough to understand what they read and answer questions,
* Women who did not want to participate in the study were not included in the sample.

Max Age: 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 352 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | initial, 1st, 1st, 3rd, 6th months and 1 year later
  The FSFI total score ranges from 2 to 36 and the FSFI total score indicates the general status of sexual function.35 The FSFI cut-off value is 26.55. A score of ≤26.55 defines sexual dysfunction and >26.55 defines normal sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No